CLINICAL TRIAL: NCT01598766
Title: General Investigational Protocol for EXCELART VANTAGE ZGV/XGV/AGV/ ATLAS/XGV/ZGV TITAN/XGV VANTAGE TITAN 3T
Brief Title: General Investigative MRI Protocol
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Toshiba America Medical Systems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 05069
Record Dates: First submitted 2012-05-11; First posted 2012-05-15 (Estimated); Last update posted 2013-02-05 (Estimated); Status verified 2013-02

CONDITIONS: Multiple MRI Exams, Including; Cardiac; Abdominal; Lumbar; Neck; Pelvis

ARMS (1):
- Diagnostic Coil (Experimental): This coil is a lightweight, flexible coil which can be used for many pediatric MRI exams
  Interventions: Device: 16 Channel SPEEDER Flex Coil

INTERVENTIONS:
Device: 16 Channel SPEEDER Flex Coil — This is a 16 element MRI coil, flexible, lightweight. Multiple uses.

SUMMARY:
This study is a feasibility study to evaluate new technology to improve the MRI experience, with coils, sequences and software. Patients from the Principle Investigator's exam schedule are given the opportunity to participate in this study is their MRI exam is appropriate for the specific coil, sequence or software being evaluated. If they agree, they can receive their MRI exam with the new coil, sequence or software instead of the standard one.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients that are scheduled for a clinically necessary MRI exam provided the subject meets the criteria of the department MRI screening procedure and their study is appropriate for the use of the 4 Channel Flex SPEEDER coil of the 16 Channel Metaflex SPEEDER coil.

Exclusion Criteria:

* Any contraindication to MRI procedures

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-05; Primary Completion 2013-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
16 Channel Flex Coil | May 2012-May 2013
  The 16 Channel Flex Coil will be evaluated for how well it performs on pediatric patients.

SECONDARY OUTCOMES:
8 Channel Value Breast Coil | 6 months
  clinical evaluation to determine if an 8 channel mri breast coil meets industry standards.

CONTACTS AND LOCATIONS:
Overall Officials: Mark L Winkler, MD, Principal Investigator — Steinberg Diagnostic Medical Imaging
Locations (1):
- Steinberg Diagnostic Medical Imaging, Henderson, Nevada, United States